CLINICAL TRIAL: NCT06113991
Title: Retrospective Multicenter Case-control Study Comparing Chronic Beryllium Disease to Pulmonary Sarcoidosis
Brief Title: Study Comparing Chronic Beryllium Disease to Pulmonary Sarcoidosis
Acronym: BERYSARC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230386
Record Dates: First submitted 2023-06-06; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Sarcoidosis; Chronic Beryllium Disease
MeSH Terms: conditions — Sarcoidosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without professional exposure to beryllium: Patients without professional exposure to beryllium
- Patients with chronic pulmonary berylliosis: Patients with chronic pulmonary berylliosis

SUMMARY:
Inhalation of beryllium can induce specific sensitization and diffuse pulmonary granulomatosis called chronic beryllium disease (CBD). The clinical, radiographic, and anatomopathological features of CBD are very similar to those of sarcoidosis, another granulomatosis, making its diagnosis difficult. In addition, the progression of CBD is poorly understood. The investigators hypothesis is that there are specific clinical, biological, anatomopathological, and radiological presentation specificities of CBD, as well as a worse prognosis compared to pulmonary sarcoidosis.

DETAILED DESCRIPTION:
Inhalation of beryllium can induce specific sensitization and diffuse pulmonary granulomatosis called chronic beryllium disease (CBD). The clinical, radiographic, and anatomopathological features of CBD are very similar to those of sarcoidosis, another granulomatosis, making its diagnosis difficult. In addition, the progression of CBD is poorly understood . The investigators hypothesis is that there are specific clinical, biological, anatomopathological, and radiological presentation specificities of CBD, as well as a worse prognosis compared to pulmonary sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Sufficiently documented medical record.
* Informed patients who did not object to participating in the research, or for deceased patients, did not object to the use of their data.
* Cases: Patients followed for confirmed chronic beryllium disease by expert teams based on the ATS 2014 criteria, i.e., a history of exposure to beryllium, positivity of two abnormal lymphocyte proliferation tests (LPT) in blood and/or an abnormal LPT in bronchoalveolar lavage, granuloma found in pulmonary biopsy associated by compatible clinical, radiological or spirometric abnormalities.
* Controls: Patients followed for sarcoidosis according to the ATS/ERS/WASOG criteria, i.e., (i) a compatible presentation, (ii) the presence of non-necrotizing granulomatosis in one or more tissues (except Löfgren's syndrome or Heerfordt syndrome), (iii) and exclusion of alternative causes of granulomatous diseases with pulmonary parenchymal involvement on thoracic CT and/or chest radiography.
* Controls: without occupational exposure to beryllium.

Exclusion Criteria:

* Patients under trustee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic beryllium disease compared to pulmonary sarcoidosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-12-14 (Estimated)

PRIMARY OUTCOMES:
The phenotypic profile at inclusion will be based on clinical data | baseline
  symptoms at diagnosis
The phenotypic profile at inclusion will be based on clinical data | baseline
  general signs(number and type of organs affected)
The phenotypic profile at inclusion will be based on biological data | baseline
  serum angiotensin-converting enzyme assay (hydrolysis of one micromole of substrate per minute)
The phenotypic profile at inclusion will be based on biological data | baseline
  blood calcium(mmol/L)
The phenotypic profile at inclusion will be based on biological data | baseline
  calciuria (mmol/kg/J)
The phenotypic profile at inclusion will be based on biological data | baseline
  blood lymphocytes(mm3)
The phenotypic profile at inclusion will be based on biological data | baseline
  gamma globulinemia (g/L)
The phenotypic profile at inclusion will be based on functional data | baseline
  extra-functional explorations with measurement in absolute value and as a percentage of the theoretical value of total lung capacity (L)
The phenotypic profile at inclusion will be based on functional data | baseline
  residual volume (%)
The phenotypic profile at inclusion will be based on functional data | baseline
  forced vital capacity (L)
The phenotypic profile at inclusion will be based on functional data | baseline
  maximum exhaled volume (L)
The phenotypic profile at inclusion will be based on functional data | baseline
  Tiffeneau (%)
The phenotypic profile at inclusion will be based on functional data | baseline
  carbon monoxide diffusion capacity (%)
The phenotypic profile at inclusion will be based on functional data | baseline
  transfer coefficient (%)
The phenotypic profile at inclusion will be based on functional data | baseline
  6-minute walk test (m)
The phenotypic profile at inclusion will be based on radiological data | baseline
  extent and description on chest CT of elementary lesions activity lesions (mm)
The phenotypic profile at inclusion will be based on radiological data | baseline
  fibrosis patterns (absence/presence)
The phenotypic profile at inclusion will be based on radiological data | baseline
  signs of pulmonary hypertension (absence/presence)

SECONDARY OUTCOMES:
Survival without transplantation | From date of baseline until the date of death,or date of lung transplantation or date of last visit whichever came first
  Survival without transplantation will be measured from the date of inclusion until death and/or lung transplantation, or the date of last follow-up.
The occurrence of comorbidities and complications related to the disease and to treatment | baseline
  The occurrence of comorbidities will correspond to the presence of comorbidities (smoking, alcoholism, obesity, diabetes, hypertension, other medical history)
Therapeutic management | baseline
  Therapeutic management will be studied by immediate indication of treatment
Psycho-social consequences | baseline and last visit in 2022
  Psycho-social consequences will be evaluated by the number of sick leaves, the existence of professional reclassification, and the number of hospitalizations
Respiratory functional evolution | baseline and last visit in 2022
  Respiratory functional evolution will correspond to the absolute variation of the respiratory function parameters extra-functional explorations with measurement in absolute value and as a percentage of the theoretical value of total lung capacity, residual volume, forced vital capacity, maximum exhaled volume, Tiffeneau, carbon monoxide diffusion capacity, transfer coefficient, 6-minute walk test, PaO2, PaCO2
CT scan evolution | last visit in 2022
  CT scan evolution will study the data from the latest available thoracic CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- 001 - Service Pneumologie, Bobigny, Avicenne, France